CLINICAL TRIAL: NCT04371094
Title: Comparison Between Using Glidescope With Stylet Technique and With Bougie Technique on the Incidence and Severity of Postoperative Sore Throat Development
Brief Title: Sore Throat After Intubation Using Glidescope With Stylet and Bougie
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Abdelrhman Alshawadfy, Lecturer of anesthesia and intensive care, Suez Canal University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: Glidescope and sore throat
Record Dates: First submitted 2020-04-27; First posted 2020-05-01 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Postoperative Sore Throat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- stylet (Active Comparator): The stylet is a device that is put inside the endotracheal tube to facilitate its insertion into the trachea
  Interventions: Device: a device to facilitate endotracheal intubation
- bougie (Active Comparator): The bougie is a device that is inserted into the trachea and an endotracheal tube is loaded over it and is slide into the trachea
  Interventions: Device: a device to facilitate endotracheal intubation

INTERVENTIONS:
Device: a device to facilitate endotracheal intubation — a device to facilitate endotracheal intubation

SUMMARY:
This is a prospective double-blinded clinical trial aiming to compare the incidence and severity of sore throat after laparoscopic cholecystectomy when using two different techniques of intubation using glidescope

DETAILED DESCRIPTION:
The first technique is loading the endotracheal tube on a stylet the second technique is sliding the endotracheal tube over a bogie that is dragged into the trachea at both techniques, the investigators are using glidescope

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II UNDERGOING LAPAROSCOPIC CHOLECYSTECTOMY UNDER GA

Exclusion Criteria:

* ANTICIPATED DIFFICULT INTUBATION

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
postoperative sore throat (POST) | IMMEDIATELY POSTOPERATIVE AND 2 HORSE LATER
  report severity of postoperative sore throat and CHANGES that could occur later on

SECONDARY OUTCOMES:
postoperative sore throat (POST) | immediately postoperative at recovery room
  INCIDENCE of postoperative sore throat

CONTACTS AND LOCATIONS:
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
STILL WORKING ON